CLINICAL TRIAL: NCT02244840
Title: The Effects of Electronic Bidet on Anal Resting Pressure, Compared to Conventional Sitz Bath in Normal Healthy Volunteers
Brief Title: Anal Resting Pressure After Bidet, Compared to Sitz Bath
Acronym: Bidet(2)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Coway Research and Development Center (Unknown)
Responsible Party: Principal Investigator, Kyu Joo Park, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0620113700
Record Dates: First submitted 2014-09-16; First posted 2014-09-19 (Estimated); Results first posted 2014-10-03 (Estimated); Last update posted 2014-10-03 (Estimated); Status verified 2014-09

CONDITIONS: Anorectal Disorders
Keywords: Bidet, Sitz bath, Anal resting pressure
MeSH Terms: conditions — Rectal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Electronic bidet and sitz bath (Experimental): Electronic bidet for 3 minutes and sitz bath for 3 minutes, at another day, for each subject
  Interventions: Device: Electronic bidet; Device: Sitz bath

INTERVENTIONS:
Device: Electronic bidet — commercial electronic bidet
Device: Sitz bath — Conventional sitz bath

SUMMARY:
Sitz bath is conventional and empirical remedy and commonly recommended for non-operative treatment of various anal diseases. However, as there was no substitute for sitz bath until now, the patients have to accept the inconvenience for treatment of their diseases.

Electronic bidet is used with convenience as automatic device for cleansing the perineal area, especially after defecation. The similarity of contacting water to perineal area, clinical use of electronic bidet has been suggested for treatment of anal diseases. However, there had been few reports of clinical use of electronic bidet.

Investigators performed the study to evaluate the effects of electronic bidet on anal resting pressure, compared to conventional warm sitz bath in normal healthy volunteers.

DETAILED DESCRIPTION:
Baseline Anorectal Manometry

The Subjects underwent a digital rectal examination and baseline anorectal manometry in the lateral decubitus position using a device from Dynacompact (Menfis Biomedica Corp., Bologna, Italy) using an 8 channel polyvinyl (PVC) catheter with the measuring orifices oriented radially. Resting and maximal pressure in the anal canal were measured by pulling the catheter out of the anorectum at a speed of 0.5 mm/sec (the 'rapid pull through' technique)

Recordings of Anal Resting Pressure on Electronic Bidet and Sitz Bath

The subjects underwent clinical experiments for recordings of anal resting pressure changes using the electronic bidet and taking the sitz bath. For the measurement of effects of electronic bidet on anal resting pressure, a different manometry catheter (8 spirally arranged channels, 0.5 cm apart) was inserted into the anal canal placing the upper channels (channels No. 1-2) with a temperature probe in the rectum and the lower channels (channel No. 3-8) in the anal canal. The catheter was fixed in the buttock area using waterproof tape and subjects sat on a toilet equipped with an electronic bidet (Coway Corp, Seoul, Korea). After anal resting pressure had stabilized at the sitting position, anal resting pressure at high pressure zone (HPZ) was checked as control value to measure the change of anal resting pressure. The anal high pressure zone (HPZ) was defined as the channel representing the highest pressure within the anal canal for each subject. The pressures while sitting were adjusted for gravity. A water flow of the electronic bidet was applied to the anus for 3 minute. We designed the new water flow system of the electronic bidet, which was fountain type with very low force (10mN), as water falls down immediately after contacting the perineal area (Fig 1A). Before applying the water flow, mist type of water particles was sprayed for a few seconds for gentle contact with water first. The water used in the electronic bidet was a tap water of warm temperature about 38 degree celsius. Anal resting pressure at the channel of HPZ was checked at 1, 2 and 3 minutes after using the electronic bidet and percentage of anal resting pressure was calculated with compared to control value checked before using the electronic bidet. Maximum and minimum pressures in the HPZ during application of the electronic bidet were noted.

Sitz bath was also undergone at another day. After insertion of catheter, the subjects were seated on a chair with small tub filled with warm water of about 38 degree celsius and sink their buttock (Fig 1B). The measurements of anal resting pressure were similar to the electronic bidet. Anal resting pressures of HPZ were checked before and after using the electronic bidet for 3 minutes. Maximum and minimum pressures were also checked.

ELIGIBILITY:
Inclusion Criteria:

* health volunteers

Exclusion Criteria:

* anorectal disorder
* medical comorbidities
* pregnancy
* history of vaginal delivery

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Jongro-gu, South Korea

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Electronic Bidet and Sitz Bath
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Electronic Bidet and Sitz Bath
Number analyzed (Participants) | 40
Age, Continuous [Mean (Full Range); unit: years] | 30.0 [22 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 20
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 40

OUTCOME MEASURES:

1. Primary Outcome: Anal Resting Pressure Change
Description: before and after bidet/sitz bath for 3 minute
Time Frame: 3 minute
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Electronic Bidet and Sitz Bath
Number analyzed (Participants) | 40
mmHg
  Baseline Electronic bidet | 90.2 (24.6)
  Post Electronic Bidet | 71.3 (23.4)
  Baseline Sitz bath | 88.1 (16.8)
  Post Sitz Bathbath | 69.6 (19.8)

2. Secondary Outcome: Convenience
Description: Questionnaires
Time Frame: 3 minute

ADVERSE EVENTS:
Arm/Group | Electronic Bidet and Sitz Bath
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes